CLINICAL TRIAL: NCT00017810
Title: Symptom Management of HIV-related Diarrhea by Using Normal Foods: A Randomized Controlled Clinical Trial.
Brief Title: The Healthy Life Choices Project in HIV-Positive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6510; R29NR004169 (NIH)
Record Dates: First submitted 2001-06-13; First posted 2001-06-14 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Diarrhea; HIV Infections
Keywords: complementary therapies; Behavior Therapy; Diarrhea; Diet Therapy; Food; HIV Seropositivity
MeSH Terms: conditions — Diarrhea; HIV Infections; HIV Seropositivity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Condition 1: Dietary Intervention (Experimental): Patients will receive behavioral dietary intervention using normal foods.
  Interventions: Behavioral: Dietary intervention
- Condition 2 (Control): HIV Self-Care (Active Comparator): Patients will receive HIV self-care information, and be given the dietary intervention at the completion of the last study session (post study).
  Interventions: Behavioral: HIV Self-Care

INTERVENTIONS:
Behavioral: Dietary intervention — The dietary intervention focused on diarrhea management using skill-building techniques that provided subjects with knowledge and a sense of confidence about making food choices.
  Behavioral dietary intervention (Condition 1: treatment) - a low-fat, lactose-free, low insoluble fiber, high soluble fiber, and caffeine-free diet based on normal foods
  Arms: Condition 1: Dietary Intervention
Behavioral: HIV Self-Care — Standard information regarding self-care and healthy living with HIV - focused on healthy living with HIV and did not include dietary restrictions or dietary information that could affect bowel movements.
  Arms: Condition 2 (Control): HIV Self-Care

SUMMARY:
This randomized clinical trial is designed to determine the efficacy of a dietary intervention to reduce the frequency of bowel movements and improve stool consistency as compared with subjects assigned to a control group. The study enrolled HIV patients with a history of three or more episodes of diarrhea for 3 weeks or more.

The purpose of this study was to compare the efficacy of a combined behavioral dietary intervention using normal foods (Condition 1: treatment) with HIV self-care (Condition 2: control) to reduce the frequency and improve the consistency of bowel movements after 3 weeks and 24 weeks of study intervention.

DETAILED DESCRIPTION:
Thirty to fifty percent of individuals with HIV can be expected to have diarrhea at some point during their illness. Diarrhea can be a chronic condition in HIV disease wherein three or more daily episodes of loose, watery stools are experienced for 4 weeks or more. Chronic diarrhea has been associated with significant morbidity, weight loss, and severe malnutrition. Researchers have reported that patients with chronic diarrhea experience a marked decrease in quality of life in comparison with HIV patients without diarrhea.

The goal of nutrition management for patients with chronic diarrhea is to ensure that adequate caloric consumption meets the metabolic needs of such individuals and to provide symptomatic relief. HIV infection, regardless of stage, causes an increase in resting energy expenditure because of the response of the body to the viral infection. Proper nutrition management can therefore assist in preventing further nutritional imbalances.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* diagnosed with HIV or AIDS based on the Centers for Disease Control and Prevention criteria
* experienced a minimum of three episodes of loose, watery, or liquid stools in a 24-hour period for at least 3 weeks
* provide verification from their primary care provider of HIV status, chronic diarrhea history, documentation of medical evaluations completed
* laboratory confirmation that stool samples were negative for pathogens
* patients who were taking antidiarrheal agents were required to be on a stable regimen (same drug, dosage, and frequency) for at least 7 days before entry into the study and still meet diarrhea frequency and consistency criteria
* antiretroviral agents taken to manage HIV required a stable regimen (same drugs, dosage, and frequency) for at least 8 weeks before study entry
* patients were required to complete a mini-mental state examination, obtaining a score of 24 or higher

Exclusion Criteria:

* not meeting any of the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1996-09; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Anastasi, PhD, Principal Investigator — Helen F. Pettit Endowed Professor of Nursing
Locations (1):
- Columbia Univ School of Nursing / Center for AIDS Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anastasi JK, Capili B, Kim AG, McMahon D, Heitkemper MM. Symptom management of HIV-related diarrhea by using normal foods: A randomized controlled clinical trial. J Assoc Nurses AIDS Care. 2006 Mar-Apr;17(2):47-57. doi: 10.1016/j.jana.2006.01.005. PMID 16800167